CLINICAL TRIAL: NCT04589234
Title: A Phase 2 Study of Saltikva (Attenuated Salmonella Typhimurium Containing the Human Gene for Interleukin-2) in Patients With Metastatic Pancreatic Cancer
Brief Title: Saltikva for Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Salspera LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSP-20-006
Record Dates: First submitted 2020-09-23; First posted 2020-10-19 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Design and Investigational Plan: Open-label, phase II, two arm, interventional, prospective, non-randomized multiple dose study in unresectable, metastatic pancreatic cancer patients 18 years of age or older
  Subject Number: 60 (30 per arm)
  Study Duration: 24 months per patient or when the patient ceases to be administered chemotherapy; whichever comes first
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saltikva with FOLFIRINOX (Experimental): 30 patients will be enrolled to receive standard of care FOLFIRINOX with oral Salmonella-IL2 (Dose 10-9) every 2 weeks for 2 years
  Interventions: Drug: Salmonella-IL2; Drug: FOLFIRINOX Alone (Historical Controls)
- Saltikva with Gemcitabine/Abraxane (Experimental): 30 patients will be enrolled to receive standard of care Gemcitabine/Abraxane with oral Salmonella-IL2 (Dose: 10-9) every 3 weeks for 2 years
  Interventions: Drug: Salmonella-IL2; Drug: Gemcitabine/Abraxane Alone (Historical Controls)

INTERVENTIONS:
Drug: Salmonella-IL2 — Phase 2 study to determine the anti-tumor effectiveness of Salmonella-IL2 (Saltikva) with standard of care chemotherapy (either FOLFIRINOX or Gemcitabine/Abraxane) for metastatic pancreatic cancer
  Other Names: Saltikva
Drug: FOLFIRINOX Alone (Historical Controls) — We will use historical data from the literature to compare FOLFIRINOX alone against the FOLFIRINOX with Salmonella-IL2 group
  Arms: Saltikva with FOLFIRINOX
Drug: Gemcitabine/Abraxane Alone (Historical Controls) — We will use historical data from the literature to compare Gemcitabine/Abraxane alone against the Gemcitabine/Abraxane with Salmonella-IL2 group
  Arms: Saltikva with Gemcitabine/Abraxane

SUMMARY:
Objectives: Assess the efficacy of multiple dose oral administration of Saltikva, an attenuated strain of Salmonella Typhimurium expressing IL-2, in patients with metastatic pancreatic cancer on standard chemotherapy (either FOLFIRINOX or Gemcitabine/Abraxane and Saltikva).

Study Rationale: The addition of Saltikva to the standard of care regimen for Stage IV metastatic pancreatic cancer will significantly prolong the overall survival and prolong the time to disease progression.

Patient Population: unresectable, metastatic pancreatic cancer patients 18 years of age or older

DETAILED DESCRIPTION:
The study agent is Saltikva, an attenuated Salmonella Typhimurium containing the gene for human IL-2 (Salmonella-IL2). Salmonella is a human pathogen typically spread via contaminated water supplies or foodstuffs. After ingestion, these bacteria invade the intestinal mucosa and colonize the gut associated lymphoid tissues, the liver, and the spleen. If pathogenic, symptoms persist for 7 to 14 days. These organisms are thought to be facultative intracellular parasites, which can persistently infect the endothelium, kupfer cells, and parenchymal cells of the liver for up to 12 weeks. The liver is considered a 'safe-site' for Salmonella as the preferred organ of residence after infection. The carrier state is eventually eradicated by the stimulation of cell-mediated and secretory immunity. Saltikva is a Salmonella based cancer therapeutic that has been genetically altered so it is incapable of causing any disease and is unable to mutate to a wild-type form of Salmonella, thus can never become pathogenic or harm anyone. Furthermore, Saltikva has been shown to preferentially invade and colonize within solid tumor tissues at a ratio of 1,000-10,000:1 over the normal 'safe-sites' of the liver. In addition, the Salmonella of Saltikva carries the gene for a powerful anti-cancer immune stimulant, Interleukin-2. Thus, Saltikva's mode of action is to invade and colonize solid tumors after oral ingestion, release a powerful immune stimulant directly within the tumor microenvironment thus avoiding systemic side effects, and imparts an immunologic mediated cancer cell kill.

Hypothesis: The addition of Saltikva to the standard of care regimen for Stage IV metastatic pancreatic cancer will significantly prolong the overall survival and prolong the time to disease progression.

Rationale for study design Two standard of care chemotherapeutic regimens are used for pancreatic cancer, namely, FOLFIRINOX and a Gemcitabine-based regimen. Despite these regimens, the median survival from Stage 4 metastatic pancreas cancer is 11.1 and 6.8 months, respectively. Oncologists choose these regimens based on the assessment of which regimen will be tolerated by the individual patients the FOLFIRINOX regimen is significantly more toxic and not as well tolerated as a gemcitabine based regimen.

Because of the significant lethality of metastatic pancreatic cancer and numerous studies conducted world wide with the two chemotherapeutic strategies that will be used in this trial, the investigators will use historical controls as comparison to the study arms in this trial. Furthermore, because the outcomes of chemotherapy only in patients with metastatic pancreatic cancer has been well documented, the investigators do not see the need for a control arm in this study. Lastly, although the patient numbers are small, the preliminary data is quite promising, and it would be considered unethical to have a control arm in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed, unresectable metastatic pancreatic adenocarcinoma
* Measurable disease will be required
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 16 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X IULN if no liver metastasis or =< 5 X IULN if liver metastases are present
* Creatinine not to be above IULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Saltikva administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients who are on immunosuppressive medications for any reason including for autoimmune diseases, organ transplantation, or hematologic conditions such as myelodysplastic syndrome.
* Patients that require ongoing antibiotics for a prophylactic reason - for example patients with chronic or frequently recurrent urinary tract infections are placed on suppressive or prophylactic antibiotics
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar biologic composition to Saltikva.
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with Saltikva but the hyperglycemia should be well controlled before the patient enters the trial (glycosylated hemoglobin [Hba1c] < 7.5)
* Patients with current evidence of significant cardiovascular disease (New York Heart Association class III or IV cardiac disease), symptomatic congestive heart failure, dilated/hypertrophic or restrictive cardiomyopathy, myocardial infarction (within the past 6 months), unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of medications for rate control for atrial fibrillation is allowed such as calcium channel blockers and beta-blockers, if stable medication for at least last month prior to initiation of Saltikva.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible. Patients with active Hepatitis B or C infection are ineligble
* Clinically significant ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 24 months
  Survival from diagnosis to death from metastatic pancreatic cancer (months)
Progression Free Survival | 24 months
  Survival from diagnosis to progression of metastatic pancreatic cancer (months)

SECONDARY OUTCOMES:
Biological response | 24 months
  Determination of CA19-9 levels (units per millimeter)
Radiologic response | 24 months
  Degree of tumor regression as determined by serial radiologic imaging (CT Scan, PET Scan, and/or MRI - percent change of tumor(s) volume (cubic millimeters)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Principal Investigator — McGill University
Locations (1):
- Segal Cancer Centre/ Mortimer B. Davis-Jewish General Hosptial, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Batist G, Kavan P, Augustin L, Schottel J, Moradian J, Lee JT, Saltzman D. A phase 2 study of orally administered live biotherapeutic salmonella-IL2 with FOLFIRINOX for stage IV pancreatic cancer. Cancer Immunol Immunother. 2026 Jan 27;75(2):60. doi: 10.1007/s00262-026-04307-0. PMID 41591505